CLINICAL TRIAL: NCT00546897
Title: Phase II Trial of Lenalidomide in Older Patients (>/= 60 Years) With Untreated Acute Myeloid Leukemia Without Chromosome 5q Abnormalities
Brief Title: Lenalidomide in Older Patients With Acute Myeloid Leukemia Without Chromosome 5q Abnormalities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0907
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Lenalidomide 50 mg/day oral for 14 days followed by 30 days of rest. Lenalidomide 50 mg/day oral for 21 days (this is Cycle 1 and Cycle 2).
  If no progressive disease (PD) then lenalidomide 10 mg/day oral for 28 days for 12 cycles.
  Interventions: Drug: Lenalidomide
- Cohort 2 (Experimental): Cycle 1: Oral lenalidomide 50 mg/day x 28 days induction therapy. Treatment will then depend on the response to Cycle 1: if patients obtain a complete remission (CR) they will proceed to low dose lenalidomide therapy, if patients have a non-CR they will receive a second high dose cycle of lenalidomide 50 mg/day x 28 days (Cycle 2) Cycle 2 consists of lenalidomide 50mg/day x 28 days Further treatment will depend on the response to Cycle 2: if patients obtain a CR/partial remission (PR)/stable disease (SD) they will proceed to low dose lenalidomide therapy, if patients have PD they will be removed from the study.
  Low Dose Cycles: low dose lenalidomide therapy consisting of 10 mg daily for a 28 day cycle.be 1) For patients that achieve a CR, 2 cycles of low dose lenalidomide will be administered, and then patients observed off therapy. For patients with PR/SD, low dose lenalidomide will continue for a total of 6 cycles and then patients will be observed off therapy.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid; CC-5013

SUMMARY:
This study is designed to test the safety and efficacy of lenalidomide in older patients (age > 60 years) with untreated acute myeloid leukemia without chromosomal abnormalities involving 5q.

DETAILED DESCRIPTION:
The incidence of AML increases with age, and current treatment options for the older patient population with newly diagnosed AML (AML >= 60) is limited, all with poor outcomes. AML >= 60 patients are more likely to have poor-risk cytogenetics abnormalities, and many have a preceding myelodysplastic syndrome (MDS). Traditional induction chemotherapy approaches in AML with cytarabine and anthracyclines yield remissions in 45-60% of AML >= 60, however the vast majority of these patients relapse with a median survival of about 9 months. These patients are rarely candidates for potentially curative allogeneic stem cell transplantation. Many untreated AML >= 60 patients are not candidates for aggressive therapy, and those who do receive therapy have a significant induction mortality of 10-20%, and significant hematologic toxicity occurs in over 30%, with no change in overall survival compared with supportive care. AML >= 60 patients with favorable risk cytogenetics have a modest improvement in prognosis, for example with a 5 year overall survival of ~20%, compared with 0% in other cytogenetic categories. Thus, all eligible patients with AML >= 60 should be recommended a clinical trial, regardless of whether they would be offered generally ineffective traditional induction chemotherapy. More effective and less toxic therapies are needed for the treatment of AML in this older patient population, indeed the preferred first line therapy in the national cancer center network (NCCN) guidelines for AML is a clinical trial.

In trials of lenalidomide in patients with MDS the dose of lenalidomide has been reduced for myelotoxicity and/or thrombocytopenia. However, current paradigms for the therapy of acute myeloid leukemia are based on using high doses of myelosuppressive chemotherapy and supporting the patient through a 4-5 weeks period of neutropenia/thrombocytopenia in an attempt to eliminate the malignant clone. Based on its efficacy in the related myeloid disorder MDS, and the close relationship between MDS and AML in patients > 60, this trial employs the same paradigm of myelosuppressive therapy using high dose lenalidomide instead of chemotherapy. Importantly, within the MDS trials using low doses of lenalidomide, responses were observed in 3/9 (33%) of patients with excess blasts (RAEB/RAEB-t), which are now classified as evolving into AML or AML. This suggests that the therapeutic effect of lenalidomide occurs in the setting of a large percentage of blasts, such as AML, although the dose and schedule of lenalidomide administration is different. The response of AML >= 60 patients to the proposed high dose lenalidomide regimen is unknown. Following high dose lenalidomide, in those patients that have a response, we propose using a lower dose maintenance strategy similar to the FDA approved dosing for MDS. The maintenance phase will include standard dose reductions for unacceptable toxicities.

ELIGIBILITY:
Inclusion Criteria:

* AML, de novo, secondary to prior therapy, or transformed from MDS, as defined by the International Working Group (except acute promyelocytic leukemia (AML M3). Patients must not have abnormalities of chromosome 5q as assessed by routine cytogenetics or FISH. Diagnosis of AML by WHO criteria (≥20% blasts) is determined by CBC, bone marrow assessment, and immunophenotypic analysis performed within 2 weeks of study enrollment.
* Intermediate or poor-risk cytogenetics as defined by SWOG criteria
* Age ≥ 60 years at the time of signing the informed consent form.
* Understand and voluntarily sign an informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* No previous treatment for AML, however hydroxyurea, steroids, and leukopheresis are allowed
* ECOG performance status of ≤ 2 at study entry.
* Life expectancy > 2 months
* Adequate organ function as defined by:
* Serum creatinine ≤ 1.5X institution upper limit of normal (ULN)
* Total bilirubin ≤ 2.0 mg/dL
* AST (SGOT) and ALT (SGPT) ≤ 5 x ULN
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.

Exclusion Criteria:

* Received prior treatment for AML
* Favorable risk cytogenetic abnormalities as defined by SWOG criteria (http://www.bloodjournal.org/cgi/content/abstract/96/13/4075) that include: inv(16)/t(16;16)/del(16q), t(15;17) with/without secondary aberrations, t(8;21) lacking del(9q) or complex karyotype (16). Prior to enrollment, FISH, molecular studies or routine cytogenetics must be completed to rule out these cytogenetic abnormalities.
* Known CNS leukemia
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 30 days of enrollment.
* Known hypersensitivity to thalidomide.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-02; Primary Completion 2010-06 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] List A, Kurtin S, Roe DJ, Buresh A, Mahadevan D, Fuchs D, Rimsza L, Heaton R, Knight R, Zeldis JB. Efficacy of lenalidomide in myelodysplastic syndromes. N Engl J Med. 2005 Feb 10;352(6):549-57. doi: 10.1056/NEJMoa041668. PMID 15703420
- [Background] List, AF, G Dewald, J Bennett, et al. 2005. Hematologic and Cytogenetic (CTG) Response to Lenalidomide (CC-5013) in Patients with Transfusion-Dependent (TD) Myelodysplastic Syndrome (MDS) and Chromosome 5q31.1 Deletion: Results of the Multicenter MDS-003 Study. In ASCO, Orlando, FL.
- [Derived] Bansal D, Vij K, Chang GS, Miller CA, DiPersio JF, Vij R, Heath SE, Westervelt P, Welch JS, Fehniger TA. Lenalidomide results in a durable complete remission in acute myeloid leukemia accompanied by persistence of somatic mutations and a T-cell infiltrate in the bone marrow. Haematologica. 2018 Jun;103(6):e270-e273. doi: 10.3324/haematol.2017.184168. Epub 2018 Mar 22. No abstract available. PMID 29567774
- [Derived] Fehniger TA, Uy GL, Trinkaus K, Nelson AD, Demland J, Abboud CN, Cashen AF, Stockerl-Goldstein KE, Westervelt P, DiPersio JF, Vij R. A phase 2 study of high-dose lenalidomide as initial therapy for older patients with acute myeloid leukemia. Blood. 2011 Feb 10;117(6):1828-33. doi: 10.1182/blood-2010-07-297143. Epub 2010 Nov 4. PMID 21051557
- [Derived] Fehniger TA, Byrd JC, Marcucci G, Abboud CN, Kefauver C, Payton JE, Vij R, Blum W. Single-agent lenalidomide induces complete remission of acute myeloid leukemia in patients with isolated trisomy 13. Blood. 2009 Jan 29;113(5):1002-5. doi: 10.1182/blood-2008-04-152678. Epub 2008 Sep 29. PMID 18824593
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 02/02/2007 and closed to participant enrollment on 03/04/2009.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 15 | 33
Completed | 15 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 15 | 33 | 48
Age, Continuous [Median (Full Range); unit: years] | 71 [60 to 86] | 71 [60 to 88] | 71 [60 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 16
  Male | 11 | 21 | 32
Region of Enrollment [Number; unit: participants]
  United States | 15 | 33 | 48
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — * 0 Fully active, able to carry on all pre-disease performance without restriction.
  * 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  * 2 Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  * 3 Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  * 4 Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  * 5 Dead
  participants
    0 | 10 | 16 | 26
    1 | 4 | 13 | 17
    2 | 1 | 4 | 5
Cytogenetic Risk Category [Number; unit: participants]
  Intermediate | 13 | 18 | 31
  Unfavorable | 2 | 13 | 15
  Unknown | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate (CRm + CRi + CRc)
Description: CRm = Defined as morphologic leukemia-free state, including <5% blasts in BM aspirate with marrow spicules and a count of > 200 nucleated cells and no blasts with Auer rods, no persistent extramedullary disease, ANC > 1000/uL, platelet count >100,000/uL. Patient must be independent of transfusions for a minimum of 1 week before each marrow assessment. There is no duration requirement for this designation.
  CRi = Defined as CR with the exception of neutropenia <1000/uL or thrombocytopenia <100,000/ul.
  Cytogenetic complete remission (CRc): Only patients with an identified cytogenetic abnormality may receive this designation. Defines as a morphologic complete remission plus reversion to a normal karyotype (no clonal abnormalities detected in a minimum of 20 mitotic cells).
Time Frame: After 2 cycles of low dose lenalidomide (approximately Day 113 for Cohort 1 and approximately Day 104 for Cohort 2)
Population: 9 out of 15 participants did not receive the two low dose cycles of lenalidomide in Cohort 1.
  23 out of 33 participants did not receive the two low dose cycles of lenalidomide in Cohort 2.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 10
participants
  CRm | 0 | 3
  CRi | 0 | 4
  CRc | 1 | 3

2. Secondary Outcome: Safety and Tolerability (Removal From Study Due to Adverse Events)
Description: Toxicity will be scored using CTCAE Version 3.0 for toxicity and adverse event reporting
Time Frame: 4 weeks after last dose of study drug [median duration of therapy was 65 days (range, 3-413 days)]
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 15 | 33
participants | 1 | 8

3. Secondary Outcome: Response Rate (RR)
Description: RR = as patients obtaining any response (CRm + CRc +CRi + PR).
  CRm = Defined as morphologic leukemia-free state, including <5% blasts in BM aspirate with marrow spicules and a count of > 200 nucleated cells and no blasts with Auer rods, no persistent extramedullary disease, ANC > 1000/uL, platelet count > 100,000/uL. Patient must be independent of transfusions for a minimum of 1 week before each marrow assessment. There is no duration requirement for this designation.
  CRc = Cytogenetic complete remission (CRc): Only patients with an identified cytogenetic abnormality may receive this designation. Defines as a morphologic complete remission plus reversion to a normal karyotype (no clonal abnormalities detected in a minimum of 20 mitotic cells).
  Morphologic complete remission with incomplete blood count recovery (CRi): Defined as CR with the exception of neutropenia <1000/uL or thrombocytopenia <100,000/ul.
  Partial remission (PR): Requires
Time Frame: After 2 cycles of low dose lenalidomide (approximately Day 113 for Cohort 1 and approximately Day 104 for Cohort 2)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 10
participants
  CRm | 0 | 3
  CRc | 1 | 3
  CRi | 0 | 4
  PR | 1 | 0

4. Secondary Outcome: Morphologic Leukemia Free State
Description: Morphologic leukemia-free state: Defined as < 5% blasts on the BM aspirate with spicules and a count of > 200 nucleated cells and no blasts with Auer rods, and no persistent extramedullary disease.
Time Frame: After 2 cycles of low dose lenalidomide (approximately Day 113 for Cohort 1 and approximately Day 104 for Cohort 2)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 10
participants | 1 | 10

5. Secondary Outcome: Morphologic Complete Remission Rate (CRm)
Description: CRm = Defined as morphologic leukemia-free state, including <5% blasts in BM aspirate with marrow spicules and a count of > 200 nucleated cells and no blasts with Auer rods, no persistent extramedullary disease, ANC > 1000/uL, platelet count >100,000/uL. Patient must be independent of transfusions for a minimum of 1 week before each marrow assessment. There is no duration requirement for this designation.
Time Frame: After 2 cycles of low dose lenalidomide (approximately Day 113 for Cohort 1 and approximately Day 104 for Cohort 2)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 10
participants | 0 | 3

6. Secondary Outcome: Cytogenetics CR Rate (CRc)
Description: Cytogenetic complete remission (CRc): Only patients with an identified cytogenetic abnormality may receive this designation. Defines as a morphologic complete remission plus reversion to a normal karyotype (no clonal abnormalities detected in a minimum of 20 mitotic cells).
Time Frame: After 2 cycles of low dose lenalidomide (approximately Day 113 for Cohort 1 and approximately Day 104 for Cohort 2)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 10
participants | 1 | 3

7. Secondary Outcome: CR With Complete Blood Counts (CRi) Rate
Description: CRi = Defined as CR with the exception of neutropenia <1000/uL or thrombocytopenia <100,000/ul.
Time Frame: After 2 cycles of low dose lenalidomide (approximately Day 113 for Cohort 1 and approximately Day 104 for Cohort 2)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 10
participants | 0 | 4

8. Secondary Outcome: Partial Remission Rate (PR)
Description: Partial remission (PR): Requires that the criteria for complete remission be met with the following exceptions: decrease of >50% in the percentage of blasts to 5-25% in the BM aspirate. A value of < 5% blasts in BM with Auer rods is also considered a partial remission.
Time Frame: After 2 cycles of low dose lenalidomide (approximately Day 113 for Cohort 1 and approximately Day 104 for Cohort 2)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 10
participants | 1 | 0

9. Secondary Outcome: Overall Survival (OS)
Description: Overall survival: Defined as the date of first dose of study drug to the date of death from any cause.
Time Frame: 2 years
Population: Participants in Cohort 1 were not analyzed for overall survival because it was determined the treatment design did not work. 8 out of 15 participants did not receive the 2 high dose lenalidomide cycles and 9 out of 15 participants did not receive any of the low dose lenalidomide cycles due to progressive disease.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 33
months |  | 4 [3 to 9]

10. Secondary Outcome: Event Free Survival (EFS)
Description: Event free survival: Defined as the interval from the date of first dose of study drug to date of treatment failure, recurrence, or death due to any cause.
Time Frame: 2 years
Population: Event free survival was not analyzed. Progression free survival was analyzed instead.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) denotes the chances of staying free of disease progression for a group of individuals suffering from a cancer after a particular treatment. It is the percentage of individuals in the group whose disease is likely to remain stable (and not show signs of progression) after a specified duration of time. Progression-free survival rates are an indication of how effective a particular treatment is.
Time Frame: 2 years
Population: Participants in Cohort 1 were not analyzed for progression-free survival because it was determined the treatment design did not work. 8 out of 15 participants did not receive the 2 high dose lenalidomide cycles and 9 out of 15 participants did not receive any of the low dose lenalidomide cycles due to progressive disease.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 33
months |  | 2 [2 to 3]

12. Secondary Outcome: Relapse Free Survival (RFS) for Complete Responders
Description: This is determined only for patients achieving a complete remission. Defined as the interval from the date of first documentation of a leukemia free state to date of recurrence or death due to any cause.
Time Frame: 2 years
Population: Participants in Cohort 1 were not analyzed for relapse free survival because it was determined the treatment design did not work. 8 out of 15 participants did not receive the 2 high dose lenalidomide cycles and 9 out of 15 participants did not receive any of the low dose lenalidomide cycles due to progressive disease.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 10
months |  | 10 [2 to NA] — NA = this is NE (not estimated). The upper bound of the 95% confidence interval was not estimable using the Kaplan-Meier survival curve

13. Secondary Outcome: Duration of CR for Complete Responders
Description: Duration of remission: Defined as the interval from the date complete remission is documented to the date of recurrence
Time Frame: 2 years
Population: Participants in Cohort 1 were not analyzed for duration of remission because it was determined the treatment design did not work. 8 out of 15 participants did not receive the 2 high dose lenalidomide cycles and 9 out of 15 participants did not receive any of the low dose lenalidomide cycles due to progressive disease.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 10
months |  | 10 [1 to 17]

14. Secondary Outcome: Changes in NK Cell Number and Function
Description: Peripheral blood mononuclear cells (PBMC) will be viably cryopreserved from patients at baseline (pre-therapy, newly diagnosed AML), during lenalidomide therapy, and posttherapy. Following sample collection, PBMC will be thawed, and flow cytometry will be performed to assess NK cell number (CD56+CD3-), subsets, and phenotype utilizing the Siteman Cancer Center Flow Cytometry / Cell Sorting Core. In addition, NK cell function will be assessed in flow based killing assays using PBMC (containing NK cells) as effectors and NK sensitive cell lines (K562) and/or autologous leukemic blasts as target cells. Thus, analyzing these parameters in patients before, during, and after therapy will provide a comprehensive evaluation of the ability of lenalidomide to modulate NK cells in patients in vivo.
Time Frame: Baseline, during therapy, and posttherapy
Population: This outcome was not analyzed for either Cohort due to number of samples collected.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Gene Expression Profiles of Bone Marrow and Peripheral Blood
Description: RNA will be made from total bone marrow cells for labeling and evaluations by RNA profiling. Cellular RNA and corresponding biotinylated cRNA targets will be prepared and hybridized with Affymetrix GeneChip® microarrays within the Multiplexed Gene Analysis SCC Core (Dr. Mark Watson, Director). Microarray data (and eventually corresponding gene sequence data) will be integrated an analyzed with state-of-the-art software packages. The pre- and post-treatment RNA profiling studies will be used as a discovery tool. Patterns of gene expression before and after lenalidomide therapy will be compared within each patient's sample to identify genes with altered expression after lenalidomide therapy. In addition, supervised algorithms will be sued to identify genes that can potentially predict clinical outcome and response to lenalidomide therapy.
Time Frame: Pre and post treatment
Population: This outcome measure was not analyzed for either Cohort due to sample collection.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Plasma Proteins Via Proteomics
Description: Proteomic analysis will be performed within the Siteman Cancer Center proteomics core on pre- and post-treatment plasma samples. This pilot proteomic study will identify candidate proteins of interest with altered expression after treatment with lenalidomide. This approach will provide an unbiased method to assess global changes in serum proteins following lenalidomide therapy.
Time Frame: Pre and post treatment
Population: This outcome was not analyzed for either Cohort due to sample collection.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment until 30 days following the completion of treatment. Cohort 1 median duration of treatment was 65 days (5-530). Cohort 2 median duration of treatment was 65 days (3-413).
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 10/15 | 25/33
Other Adverse Events (participants affected / at risk) | 15/15 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=15) | Cohort 2 (N=33)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 12
Pneumonia (Infections and infestations) | 2 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 0
Death due to progressive disease (General disorders) | 3 | 6
Staph hominis bacteremia infection (Infections and infestations) | 1 | 0
Catheter line infection (Infections and infestations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dehydration (Gastrointestinal disorders) | 1 | 2
Opportunistic fungal infection - death (Infections and infestations) | 1 | 0
Lower extremity weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Fatigue (General disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Syncope (Cardiac disorders) | 0 | 3
Petichae (Skin and subcutaneous tissue disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Death due to CNS hemorrhage (Nervous system disorders) | 1 | 0
Gram-cocci infection (Infections and infestations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypernatremia (Investigations) | 0 | 1
Hypokalemia (Investigations) | 0 | 1
Neutrophils (Investigations) | 0 | 2
Platelets (Investigations) | 0 | 1
Splenic infarction (Gastrointestinal disorders) | 0 | 1
Streptococcus bacteremia infection (Infections and infestations) | 0 | 1
Death due to acute renal failure (Renal and urinary disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Chest pain (Cardiac disorders) | 0 | 2
Subdural hematoma (Nervous system disorders) | 0 | 1
E. Coli infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Mucositis (Gastrointestinal disorders) | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Coryn bacterium miutissimum sepsis (Infections and infestations) | 0 | 1
Staphylcoccus epidermidis sepsis (Infections and infestations) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Mental status (Psychiatric disorders) | 0 | 1
Gram positive sepsis (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Liver dysfunction (Hepatobiliary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsil fistula (Gastrointestinal disorders) | 0 | 1
Coagulase negative staphylococcus sepsis (Infections and infestations) | 0 | 1
Cardiac ischemia (Cardiac disorders) | 0 | 1
C. difficile colitis (Gastrointestinal disorders) | 0 | 1
Upper GI hemorrhage (Gastrointestinal disorders) | 0 | 1
Lower GI hemorrhage (Gastrointestinal disorders) | 0 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=15) | Cohort 2 (N=33)
Abdominal pain (Gastrointestinal disorders) | 1 | 7
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 2
Alkaline phosphatase (Investigations) | 4 | 10
Alkylosis (Investigations) | 1 | 0
Allergic reaction/hypersensitivity (Immune system disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Back spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Bilirubin (Investigations) | 3 | 12
Biopsy site pain (Surgical and medical procedures) | 1 | 3
Blurred vision (Eye disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
CNS hemorrhage (Nervous system disorders) | 0 | 1
Cardiac ischemia (Cardiac disorders) | 0 | 2
Cardiopulmonary arrest (Cardiac disorders) | 1 | 0
Chest pain (Cardiac disorders) | 2 | 5
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Chills (General disorders) | 1 | 5
Confusion (Psychiatric disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 3 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Creatinine (Investigations) | 2 | 12
Cystitis (Renal and urinary disorders) | 0 | 1
Decubitus (Skin and subcutaneous tissue disorders) | 0 | 1
Dehydration (Gastrointestinal disorders) | 0 | 4
Dental abscess (Gastrointestinal disorders) | 0 | 1
Dental pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 12
Diverticulosis (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 13
Edema (Investigations) | 7 | 11
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Eye hemorrhage (Eye disorders) | 0 | 2
Fatigue (General disorders) | 8 | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 14
Feet pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fever (no infection) (General disorders) | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Floaters (Eye disorders) | 0 | 1
Generalized pain (General disorders) | 0 | 7
Hand pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hard palate ulcer (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 3
Hematoma (Vascular disorders) | 1 | 1
Hemoglobin (Blood and lymphatic system disorders) | 10 | 22
Hemorrhagic lesion (Vascular disorders) | 1 | 0
Hemorrhoid pain (Gastrointestinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperglycemia (Investigations) | 3 | 6
Hyperkalemia (Investigations) | 2 | 3
Hypermagnesemia (Investigations) | 1 | 1
Hypernatremia (Investigations) | 5 | 5
Hypertension (Cardiac disorders) | 0 | 6
Hyperuricemia (Investigations) | 1 | 1
Hypoalbuminemia (Investigations) | 8 | 19
Hypocalcemia (Investigations) | 12 | 21
Hypokalemia (Investigations) | 4 | 14
Hyponatremia (Investigations) | 8 | 11
Hypophosphatemia (Investigations) | 1 | 2
Hypotension (Cardiac disorders) | 1 | 6
Hypothyroidism (Endocrine disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 6
INR (Investigations) | 2 | 0
Incontinence - anal (Gastrointestinal disorders) | 1 | 5
Infection w/neutropenia - cellulitis (Infections and infestations) | 0 | 1
Infection w/neutropenia - clostridium difficile (Infections and infestations) | 0 | 1
Infection w/neutropenia - enterococcus faecium (Infections and infestations) | 0 | 1
Infection w/neutropenia - escheria coli (Infections and infestations) | 0 | 1
Infection w/neutropenia - oral candidiasis (Infections and infestations) | 0 | 2
Infection w/neutropenia - parainfluenza (Infections and infestations) | 0 | 1
Infection w/neutropenia - pneumonia (Infections and infestations) | 3 | 11
Infection w/neutropenia - polymicrobial sepsis (Infections and infestations) | 0 | 1
Infection w/neutropenia - stapphylococcus (Infections and infestations) | 2 | 5
Infection w/neutropenia - unspecified (Infections and infestations) | 2 | 0
Infection w/neutropenia - upper respiratory (Infections and infestations) | 1 | 1
Infection w/neutropenia - urinary tract (Infections and infestations) | 0 | 1
Infection w/neutropenia - vaginal (Infections and infestations) | 0 | 1
Infection w/o neutropenia - bronchitis (Infections and infestations) | 0 | 1
Infection w/o neutropenia - catheter fungemia (Infections and infestations) | 1 | 0
Infection w/o neutropenia - coagulase negative staphylococcus bacteremia (Infections and infestations) | 0 | 2
Infection w/o neutropenia - middle ear (Infections and infestations) | 1 | 0
Infection w/o neutropenia - oral candidiasis (Infections and infestations) | 0 | 1
Infection w/o neutropenia - pneumonia (Infections and infestations) | 0 | 3
Infection w/o neutropenia - upper respiratory (Infections and infestations) | 1 | 1
Inguinal hernia (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 1
Leukocytes (WBC) (Investigations) | 9 | 15
Liver dysfunction (Hepatobiliary disorders) | 0 | 1
Lower GI NOS hemorrhage (Gastrointestinal disorders) | 0 | 1
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Lymphocele (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Investigations) | 1 | 0
Mood alteration - agitation (Psychiatric disorders) | 0 | 1
Mood alteration - anxiety (Psychiatric disorders) | 0 | 2
Mood alteration - depression (Psychiatric disorders) | 1 | 1
Mucositis (Gastrointestinal disorders) | 1 | 11
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness - generalized (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle weakness - lower extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 9
Neck nodule (General disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutrophils (ANC) (Investigations) | 8 | 11
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Palpitations (Cardiac disorders) | 1 | 0
Peridontal - mandible swelling (Gastrointestinal disorders) | 1 | 0
Periodontal - poor dentition (Gastrointestinal disorders) | 1 | 2
Petechiae (Vascular disorders) | 2 | 6
Platelets (Investigations) | 12 | 25
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Progressive disease (General disorders) | 2 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 1
Psychosis - hallucinations (Psychiatric disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 18
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rib pain (Musculoskeletal and connective tissue disorders) | 0 | 2
SGOT (AST) (Investigations) | 8 | 12
SGPT (ALT) (Investigations) | 12 | 14
Sensory neuropathy (Nervous system disorders) | 0 | 4
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Sinus drainage (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 7
Sinusitis (Infections and infestations) | 0 | 2
Skin sore (Skin and subcutaneous tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Splenic infarction (Gastrointestinal disorders) | 0 | 1
Supraventricular arrhythmia (Cardiac disorders) | 1 | 0
Sweating (General disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 4
Taste alteration (Gastrointestinal disorders) | 0 | 2
Throat pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Thrombosis (Vascular disorders) | 0 | 2
Tingling in extremities (Nervous system disorders) | 0 | 2
Tonsil fistula (Gastrointestinal disorders) | 0 | 1
Tremors (Nervous system disorders) | 0 | 1
Upper extremity pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 4
Vasculitis (Vascular disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 6
Weight loss (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes